CLINICAL TRIAL: NCT03319433
Title: Prediction of Hypotension Using Perfusion Index Following Spinal Anesthesia in Lower Segment Caesarean Section
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Paropakar Maternity and Women's Hospital (Other)
Responsible Party: Principal Investigator, Achyut Sharma, Dr., Paropakar Maternity and Women's Hospital
Other Study IDs: ParopakarMWH
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Spinal; Hypotension; Perfusion Index
Keywords: spinal hypotension; perfusion index; caesarean section
MeSH Terms: conditions — Hypotension | interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I (Perfusion Index <3.5): Those parturient with perfusion index <3.5 when baseline monitors are attached while the patient is being prepared for surgery.
  Interventions: Device: Perfusion Index
- Group II (Perfusion index >3.5): Those parturient with perfusion index >3.5 when baseline monitors are attached while the patient is being prepared for surgery.
  Interventions: Device: Perfusion Index

INTERVENTIONS:
Device: Perfusion Index — Use of non-invasive pulse oximeter to determine perfusion index

SUMMARY:
Spinal anesthesia for caesarean section is invariably associated with variable degree of hypotension. Hypotension that occurs may be detrimental to various organ system due to inadequate perfusion. Various methods and agents have been tried in order to address this problem. However, this calamity is far from over.

Perfusion index is one such attempt to address the problem of hypotension by predicting which group of parturient may develop hypotension. This is a type of non-invasive method of assessing the relative vascular tone with the use of pulse oximeter which calculates the ration of pulsatile versus the non-pulsatile component of the blood flow. During normal physiological changes in pregnancy, there is relative loss of vascular tone which predisposes this group of patient to sudden development of hypotension after the sympathetic block due to spinal anesthesia.

Thus, the aim of the study is to use the non-invasive perfusion index data to predict the occurrence of hypotension in a parturient so that helps us to guide fluid and other drug therapy to address the problem of hypotension.

ELIGIBILITY:
Inclusion Criteria:

1. ASA II physical status.
2. Planned for elective LSCS
3. Gestational age >36 weeks and <41 weeks

Exclusion Criteria:

1. Patient's refusal.
2. Emergency LSCS.
3. Patient's with contraindications to spinal anesthesia
4. Patient with BMI >40, preeclampsia, placenta praevia.
5. Patients with comorbidities like cerebrovascular or cardiovascular disease, and gestational diabetes.

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Parturient presenting to Paropakar Maternity and Women's Hospital for elective caesarean section.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-08-30 (Estimated); Study Completion 2018-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension | 3 months
  compare the incidence of hypotension following SAB for LSCS in parturient with or without a high perfusion index.

SECONDARY OUTCOMES:
Perfusion index | 3 months
  To compare the perfusion index (PI) at various intervals between the two groups
Side-effects | 3 months
  To study the profile of side effects between the two groups.
Systolic blood pressure | 3 months
  To compare the systolic blood pressure (SBP) at various intervals between the two groups.
Diastolic blood pressure | 3 months
  To compare the diastolic blood pressure (DBP) at various intervals between the two groups.
Mean arterial pressure | 3 months
  To compare the mean arterial pressure (MAP) at various intervals between the two groups

REFERENCES:
- [Result] Soma-Pillay P, Nelson-Piercy C, Tolppanen H, Mebazaa A. Physiological changes in pregnancy. Cardiovasc J Afr. 2016 Mar-Apr;27(2):89-94. doi: 10.5830/CVJA-2016-021. PMID 27213856
- [Result] Chooi C, Cox JJ, Lumb RS, Middleton P, Chemali M, Emmett RS, Simmons SW, Cyna AM. Techniques for preventing hypotension during spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2017 Aug 4;8(8):CD002251. doi: 10.1002/14651858.CD002251.pub3. PMID 28976555
- [Result] Nag DS, Samaddar DP, Chatterjee A, Kumar H, Dembla A. Vasopressors in obstetric anesthesia: A current perspective. World J Clin Cases. 2015 Jan 16;3(1):58-64. doi: 10.12998/wjcc.v3.i1.58. PMID 25610851
- [Result] Duggappa DR, Lokesh M, Dixit A, Paul R, Raghavendra Rao RS, Prabha P. Perfusion index as a predictor of hypotension following spinal anaesthesia in lower segment caesarean section. Indian J Anaesth. 2017 Aug;61(8):649-654. doi: 10.4103/ija.IJA_429_16. PMID 28890560